CLINICAL TRIAL: NCT02391974
Title: Filling of Periodontal Pockets With a Commercially Available Injectable Cross-linked Hyaluronic Acid Dental Filler Versus Oral Hygiene Alone, After Scaling and Root Planing and Chlorhexidine Disinfection, for the Treatment of Periodontitis: A Single-blinded, Multi Center, Prospective, Randomized Controlled Trial
Brief Title: Efficacy and Safety of a Commercially Available Injectable Hyaluronic Acid Dental Filler for Periodontal Pockets
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teoxane SA (Industry)
Collaborators: Syneed Medidata GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-PER-1401
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Periodontitis
Keywords: Hyaluronic acid; Periodontal pockets; Periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Pocket; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PERIOSYAL FILL (Experimental): n=15
  Interventions: Device: PERIOSYAL FILL
- No treatment (untreated control) (No Intervention): n=15

INTERVENTIONS:
Device: PERIOSYAL FILL — Injection 2 weeks after standard periodontal treatment procedure on all teeth that need to be treated.
  Touch-up treatment provided at 3 and 6 weeks.
  Arms: PERIOSYAL FILL

SUMMARY:
This is a controlled, randomized, single-blinded, multicenter, prospective clinical study.

In addition to the standard periodontal treatment procedure on all teeth that need to be treated, the 4 teeth with the deepest pockets (between 4 and 6 mm) will be randomized to either PERIOSYAL® FILL and oral hygiene or oral hygiene alone.

The pocket depth will be measured at six sites around each tooth, and only the deepest pocket sites of each tooth will be taken into account.

DETAILED DESCRIPTION:
This is a controlled, randomized, single-blinded (independent Blinded Evaluator), multicenter, prospective clinical study.

Each subject will receive the standard periodontal treatment procedure on all teeth that need to be treated. The usual cares are scaling and root planing (SRP), and chlorhexidine, and instructions to oral hygiene (proper brushing techniques twice a day, proper flossing technique daily, and prevention : sugar intake, alcohol consumption, fluoride level).

Two other optional treatment sessions with SRP could be performed, if deemed necessary by the Treating Investigator. Those optional SRP session could only be performed after all study-related clinical assessement.

The pocket depth of every teeth will be measured at six sites around each tooth, and only the deepest pocket sites will be taken into account. The 4 teeth with the deepest pockets will be included in the study and randomized to either PERIOSYAL® FILL and oral hygiene or oral hygiene alone.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged between 25 and 60 years
* Patients with at least 20 natural teeth
* Patient with periodontitis confirmed by a X-ray diagnosis, and having at least 4 teeth with periodontal pockets with probing depth between 4 and 6 mm
* Willing to understand and comply with study requirements and to sign informed consent

Exclusion Criteria:

* Patient with an active smoking status
* Patient with an antibiotic therapy within the previous 4 weeks
* Need for continuous medical treatment within 2 weeks prior to enrollment
* Ongoing inflammatory state or a systemic illness that may affect the oral cavity
* Patient with hypofunction in saliva productions (e.g. Sjögren Syndrome with Xerostomia)
* History of active chronic debiliating systemic disease, including insulin or non-insulin dependent diabetes
* Patients with bleeding disorders
* History of allergies to gram positive bacterial proteins
* History of hypersensitivity and/or idiosyncrasies to any of the test compounds, e.g. hyaluronic acid or other device compounds
* History of multiple severe allergies, history of anaphylactic shock
* History of connective tissue disease (rheumatoid arthritis, scleroderma, systemic lupus erythematosus) or of any other autoimmunity disease
* History of herpetic lesion or lichen planus
* Pregnant or breast feeding women, or female subjects of childbearing potential who did not intend to practice medically acceptable method of contraception
* Participation in another clinical study in the previous 3 months

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-10 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in Pocket Probing Depth (PPD) | Pre-injection, to 12, 24 and 48 weeks after baseline
  PPD is defined as the distance from the gingival margin to the base of the gingival crevice, i.e. the bottom of the clinical pocket. PPD will be measured at six sites per tooth (DV, V, MV, DL, L, ML), using a constant-force computerized periodontal probe with a 0.2 mm precision. Only the deepest will be taken into account

SECONDARY OUTCOMES:
Change in Pocket Probing Depth (PPD) | Pre-injection, to 2, 5, 8 and 36 weeks after baseline
Change in Clinical Attachment Level (CAL) | Pre-injection, to 2, 5, 8, 12, 24, 36 and 48 weeks after baseline
  CAL is defined as the distance from the Cemento-Enamel Junction (CEJ) to the base of the probable crevice/pocket (the bottom of the clinical pocket)
Bleeding On Probing (BOP) | Pre-injection, to 2, 5, 8, 12, 24, 36 and 48 weeks after baseline
  BOP is defined as presence/absence of bleeding within 15 seconds following pocket probing
Tooth Mobility | Pre-injection, to 12, 24, 36 and 48 weeks after baseline
  Tooth Mobility will be assessed on the scale defined by Muehlemann
Plaque Index (PI) | Pre-injection, to 2, 5, 8, 12, 24, 36 and 48 weeks after baseline
  PI will be measured for each tooth using the four-point scale Silness and Löe Plaque Index
Gingival Index (GI) | Pre-injection, to 2, 5, 8, 12, 24, 36 and 48 weeks after baseline
  GI will be measured for each tooth using the four-point scale Silness and Löe Gingival Index
Oral Health-related quality of life | Pre-injection, to 12, 24, 36 and 48 weeks after baseline
  Oral Health-related quality of life is a patient reported outcome measure specifically pertaining to oral health capturing both the functional, social and psychological impacts of oral disease, assessed using the OHQoL-GE, a validated translation of the OHQoL-UK
Microbiological analysis of the 11 main periodontal pathogens | : Pre-injection, to 12, 24, 36 and 48 weeks after baseline
  Periodontal pathogens will be measured using micro-IDent plus 1/11 Hain tests, a noninvasive saliva prelevement using paper points
Physician satisfaction with the treatment | 12, 24, 36 and 48 weeks after baseline
  Satisfaction will be assessed on a 5-grade subjective symmetrical scale
Subject Satisfaction with the treatment | 12, 24, 36 and 48 weeks after baseline
  Satisfaction will be assessed on a 5-grade subjective symmetrical scale
Total volume of product injected in each of the included teeth | during each injection session
  Volume will be measured to an accuracy of 0.025 mL
Pain felt by the patient in the aera (tooth, gum) | Pre-injection, to 2, 5, 8, 12, 24, 36 and 48 weeks after baseline
  Pain will be self-assessed by the subject on each included teeth using a 100 mm Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Dental Specialist, Düsseldorf
  - Dr. Wahlmann & Partner, Edewecht
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg